CLINICAL TRIAL: NCT00950391
Title: Enhancement of Functional Recovery After Peripheral Nerve Injury With Tacrolimus
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: PI unable to secure funding for the project so study was not pursued.
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FK50600
Record Dates: First submitted 2009-07-29; First posted 2009-07-31 (Estimated); Last update posted 2018-02-13 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Nerve Injury
Keywords: peripheral nerve injury; peripheral nerve surgery; nerve repair; nerve graft
MeSH Terms: conditions — Peripheral Nerve Injuries | interventions — Tacrolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Tacrolimus (Experimental): Treatment with tacrolimus following nerve repair/reconstruction
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus — Tacrolimus 3 mg/day taken twice daily to maintain blood level of 3-6 ng/ml for duration of 1 year or less
  Other Names: FK506, Prograf

SUMMARY:
Tacrolimus (FK506) is an immunosuppressive medication that promotes organ allograft survival. It has also been shown to enhance nerve regeneration and muscle reinnervation in animals but these properties have not previously been studied in patients. Moreover, currently there is no method in clinical use to speed the rate of recovery after nerve injury. The objective of this study is to explore the ability of tacrolimus to benefit the treatment of patients with peripheral nerve injury. To minimize the morbidity of tacrolimus therapy, its phase-specific effects on nerve regeneration and muscle reinnervation will be defined in the murine model to permit further limitation of the duration of therapy. The investigators hypothesize that treatment with tacrolimus after autogenous peripheral nerve reconstruction will accelerate nerve regeneration, reduce the period of denervation and improve muscle reinnervation and recovery in patients with peripheral nerve injury.

There are 2 specific aims:

1. Determine the safety and efficacy of tacrolimus following reconstructive nerve surgery in a double-blind placebo-controlled randomized pilot clinical trial of patients with severe nerve injuries of the extremities;
2. Correlate the quality of life outcome with assessment of functional recovery after surgical reconstruction of patients with severe peripheral nerve injuries of the extremities.

ELIGIBILITY:
Inclusion Criteria:

1. have deficit of upper extremity function of MRC grade 0-2
2. are candidates for surgical reconstruction
3. are no more than 10 months after their injury
4. have no ongoing infectious or wound healing complications related to injury or previous surgery or otherwise
5. have no history of cancer or have been treated and free of cancer for at least 5 years
6. age 18-50
7. agree to participate in the study

Exclusion Criteria:

1. positive HIV or hepatitis blood test
2. recent history of cancer within the past 5 years
3. history of severe and recurrent infections (such as hidradenitis suppurativa)
4. presence of ongoing and unresolved infectious concerns related to original injury or previous surgery (such as osteomyelitis, wound infection) or otherwise
5. presence of ongoing wound healing problems related to the injury or previous surgery or otherwise
6. presence of moderate or severe liver disease as indicated by aspartate transaminase (AST), alanine transaminase (ALT), amino alkaline phosphatase, or total bilirubin levels greater than the upper limit of normal (ULN)
7. creatinine level ≥ 1.0 mg/dl or more than ULN
8. hemoglobin value of <9.0 mg/dl, a white blood cell count <3,000 cells/mm3, or platelet count <100,000 platelets/mm3
9. uncontrolled hypertension with systolic blood pressure >160 mm Hg and diastolic blood pressure >90 mm Hg at screening and baseline
10. hyperkalemia (serum K > ULN)
11. pancreatitis or diabetes mellitus (fasting blood sugar ≥ 110 mg/dl or postprandial blood sugar ≥ 160 mg/dl) or a history of these
12. heart disease or abnormal electrocardiogram (ECG) especially arrhythmia and change in ST/T or a previous history of these
13. history of serious drug hypersensitivity
14. age less than 18 or greater than 50
15. incarceration prior to or at the time of consideration for enrollment (any participant who becomes incarcerated during the course of the study will be excluded)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2014-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Functional Recovery | 1-1.5 years
Incidence of adverse events. | 1 year

SECONDARY OUTCOMES:
Recovery time. | 1.5 years
Recovery of sensation. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Thomas H Tung, MD, Principal Investigator — Washington University School of Medicine